CLINICAL TRIAL: NCT06316947
Title: Developing and Pilot Testing an Intervention to Reduce Household Shisha Smoke Exposure Within Somali Homes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMCH-2024-32723
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Shisha
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Intervention Model Description: a feasibility pilot of the new CHW-delivered intervention to reduce home shisha SHS exposure with n=15 Somali families.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Families (Experimental): Somali American families with children in the household and at least one adult using shisha at home
  Interventions: Radiation: CHW-delivered intervention

INTERVENTIONS:
Radiation: CHW-delivered intervention — WellShare CHWs will then deliver the brief, approximately 15-minute intervention to the participating parent. The new intervention components will build off existing tobacco education outreach using verbal instruction and images developed by WellShare CHWs and layer in home smoke-free rules, potential biomarker feedback about smoke exposure, and other educational intervention components that align. Additionally there will be pre and post-intervention surveys and urine samples collection for cotinine levels.

SUMMARY:
Previous qualitative research among Somali American adults in Minnesota have identified high levels of hookah or shisha (hereafter shisha) use in Somali households. Household shisha use exposes all family members, including children, to secondhand smoke (SHS) that contains toxins that can cause many different acute and chronic disease, including increased levels of several cancers such as lung, bladder, and oral cancers. Despite the high levels of shisha use, gaps in the knowledge of the risks of shisha use and how to mitigate the potential harmful health consequences of shisha use exist among Somali Americans.

This study aims to pilot test the feasibility of a newly developed CHW-delivered intervention to reduce home shisha SHS exposure with n=15 Somali families. Pre-/post-measurements of family members' (1 adult and 1 child) urine or salivary cotinine levels will be obtained along with a brief pre-/post-survey to characterize household tobacco use and the presence of home smoke-free rules.

ELIGIBILITY:
Inclusion Criteria:

Eligible families will identify as

* Somali American,
* have one or more children between 6 months and 18 years of age in the home, and
* have at least one adult who uses shisha at home. Families with other forms of tobacco use in addition to shisha use will be included.

Exclusion Criteria:

* Participation in previous qualitative study to inform intervention development
* Inability or unwillingness to provide informed consent and complete all study procedures

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 8 weeks
  number of recruited participants out of number of approached
Retention rate measure | 8 weeks
  proportion of participants who complete the 2 visits for data collection
pre-/post- survey completion rates | 8 weeks
  proportion of participants who complete the pre and post-intervention surveys
pre-/post- biospecimen completion rates | 8 weeks
  proportion of participants who complete the urine sample collection

SECONDARY OUTCOMES:
shisha use changes | 8 weeks
  Pre-/post- changes (baseline to 8 week follow-up) in the frequency of shisha use. A pre-pilot survey has been developed and will assess this outcome measure.
tobacco product use changes | 8 weeks
  Pre-/post- changes in the frequency of other tobacco product use. A pre-pilot survey has been developed and will assess this outcome measure.
smoke-free home rules | 8 weeks
  Pre-/post- changes in the presence of smoke-free home rules. A pre-pilot survey has been developed and will assess this outcome measure.
the cotinine levels of parents and children. | 8 weeks
  Pre-/post- changes in the cotinine levels of parents and children.

CONTACTS AND LOCATIONS:
Overall Officials: April Wilhelm, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States